CLINICAL TRIAL: NCT06587321
Title: The ReASSure-PC Study: A Feasibility Study of Remote Assessment of Signs and Symptoms in Palliative Care
Brief Title: Remote Assessment of Signs and Symptoms in Palliative Care
Acronym: ReASSure-PC
Status: Recruiting | Type: Observational
Sponsor: Our Lady's Hospice and Care Services (Other)
Responsible Party: Principal Investigator, Prof Andrew Davies, Professor of Palliative Medicine, Our Lady's Hospice and Care Services
Other Study IDs: RS23-078
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Palliative Care; Vital Signs; Remote Monitoring
Keywords: Remote monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Digital health interventions, including remote monitoring of patients, have been identified as a possible way to address current problems within the health service, including insufficient numbers of staff, and an increasing number of patients requiring services.

The aim of this study is to assess the feasibility of using remote monitoring for patients who are receiving palliative care and to see whether remote monitoring can improve care and outcomes for patients and their families.

Participants in this study will complete regular (daily, weekly, monthly) questionnaires online about how they are feeling. They will also be given equipment to measure their vital signs every day. The clinical team will have access to the results and be able to respond to any new problems as they arise. Patients and their carers will then complete a questionnaire at one month to assess satisfaction with the use of remote monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of advanced cancer or another life-limiting condition
* Estimated prognosis greater than 3 months
* Referred for community-based specialist palliative care
* Living in own home (or home of family carer)
* Living with a family carer

Exclusion Criteria:

* Estimated prognosis less than 3 months or more than 12 months
* Cognitive impairment - unable to provide consent / complete assessments
* Non-English speaker
* Living in care home / nursing home / hospice / community hospital
* Not living with a family carer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a diagnosis of a life-limiting condition, who are receiving care from the community palliative care team
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Completion rates of assessments | At the end of 1 month
  Number of assessments completed over the study time-frame

SECONDARY OUTCOMES:
Recruitment rate | 6 months
  The number of patients approached to take part in the study who then entered the study
Retention rate | 6 months
  The number of patients who entered and then completed the study
Acceptability | 1 month
  A patient / carer acceptability questionnaire completed at 1 month into study period
Use of community palliative care resources | 6 months
  Number of phone calls / visits / interventions participants receive
Use of GP / hospital resources | 6 months
  The number of unplanned GP visits / hospital attendances over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Power, Principal Investigator — Our Lady's Hospice & Care Services
Locations (1):
- Our Lady's Hospice & Care Services, Dublin, Dublin, Ireland